CLINICAL TRIAL: NCT05529966
Title: Comparing NGENUITY vs Conventional Microscope in a New Hydrus User
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: Alcon Research (Industry)
Responsible Party: Principal Investigator, Robert T. Chang, MD, Associate Professor of Ophthalmology, Stanford University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 66363
Record Dates: First submitted 2022-09-02; First posted 2022-09-07 (Actual); Results first posted 2025-04-08 (Actual); Last update posted 2025-04-17 (Actual); Status verified 2025-04

CONDITIONS: Glaucoma
MeSH Terms: conditions — Glaucoma

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- NGENUITY (Experimental): Research fellow participants utilize NGENUITY during micro-stent placement
  Interventions: Device: NGENUITY
- Conventional microscope (Active Comparator): Research fellow participants utilize conventional microscope during micro-stent placement
  Interventions: Device: Conventional microscope

INTERVENTIONS:
Device: NGENUITY — Device for 3-D viewing during placement of micro-stent placement.
  Arms: NGENUITY
Device: Conventional microscope — Device for stereoscopic viewing during placement of micro-stent placement.
  Arms: Conventional microscope

SUMMARY:
To compare the potential efficiency and educational value of using NGENUITY (3D camera system, FDA approved for this indication) vs the conventional microscope for Hydrus microstent placement by new users.

ELIGIBILITY:
Inclusion Criteria:

* Patients with mild to moderate primary open angle glaucoma as defined by AGS with visually significant age-related cataract undergoing uncomplicated cataract surgery and Hydrus microstent
* Either eye or both eyes may participate

Exclusion Criteria:

* Lack of patient cooperation severely affecting ability to place stent with any visualization technique
* Angle abnormalities including PAS in nasal quadrant
* Unable to properly visualize the angle due to complicated cataract surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2023-02-13 (Actual); Primary Completion 2024-03-22 (Actual); Study Completion 2024-03-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert T Chang, MD, Principal Investigator — Stanford University
Locations (1):
- Byers Eye Institute, Palo Alto, California, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 32 participants signed informed consent, 28 were randomized to either study arm.
Units Other Than Participants: Eyes
Groups:
- Conventional Microscope: Participants randomized to the use of a conventional microscope for the first eye procedure. Participants who had a procedure for their second eye were randomized again to either the conventional or NGENUITY microscope.
- NGENUITY: Participants randomized to the use of a NGENUITY microscope for the first eye procedure. Participants who had a procedure for their second eye were randomized again to either the conventional or NGENUITY microscope.
- Conventional Microscope (Re-randomized): Participants who had a procedure for their second eye were re-randomized to use of a conventional microscope for the procedure.
- NGENUITY (Re-randomized): Participants who had a procedure for their second eye were re-randomized to use of the NGENUITY microscope for the procedure.
Period: First Eye
Arm/Group | Conventional Microscope | NGENUITY | Conventional Microscope (Re-randomized) | NGENUITY (Re-randomized)
Started | 14; 14 Eyes | 14; 14 Eyes | 0; 0 Eyes | 0; 0 Eyes
Stent Placement Could Not be Performed | 1; 1 Eyes | 1; 1 Eyes | 0; 0 Eyes | 0; 0 Eyes
Had Missing Data | 1; 1 Eyes | 0; 0 Eyes | 0; 0 Eyes | 0; 0 Eyes
Evaluable for Primary and Secondary Outcome Measure Analysis | 12; 12 Eyes | 13; 13 Eyes | 0; 0 Eyes | 0; 0 Eyes
Completed | 13; 13 Eyes | 13; 13 Eyes | 0; 0 Eyes | 0; 0 Eyes
Not Completed | 1; 1 Eyes | 1; 1 Eyes | 0; 0 Eyes | 0; 0 Eyes
Period: Second Eye
Arm/Group | Conventional Microscope | NGENUITY | Conventional Microscope (Re-randomized) | NGENUITY (Re-randomized)
Started | 0; 0 Eyes | 0; 0 Eyes | 1; 1 Eyes | 3; 3 Eyes
Randomized to Use of Opposite Microscope for Second Eye Procedure | 0; 0 Eyes | 0; 0 Eyes | 1; 1 Eyes | 2; 2 Eyes
Evaluable for Primary and Secondary Outcome Measure Analysis | 0; 0 Eyes | 0; 0 Eyes | 1; 1 Eyes | 3; 3 Eyes
Completed | 0; 0 Eyes | 0; 0 Eyes | 1; 1 Eyes | 3; 3 Eyes
Not Completed | 0; 0 Eyes | 0; 0 Eyes | 0; 0 Eyes | 0; 0 Eyes

BASELINE CHARACTERISTICS:
Population: Participants/eyes evaluable for primary and secondary outcome measure analysis
Groups:
- Total: Total of all reporting groups
Arm/Group | Conventional Microscope | NGENUITY | Total
Number analyzed (Participants) | 12 | 13 | 25
Age, Continuous [Mean (Standard Deviation); unit: years] | 75.6 (8.1) | 76.1 (7.3) | 75.9 (7.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 6 | 13
  Male | 5 | 7 | 12
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 1
  Not Hispanic or Latino | 12 | 12 | 24
  Unknown or Not Reported | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian | 0 | 1 | 1
  Asian | 6 | 2 | 8
  Black | 0 | 1 | 1
  Other | 2 | 0 | 2
  White | 4 | 9 | 13
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 12 | 13 | 25

OUTCOME MEASURES:

1. Primary Outcome: Time of First Cannula in Until Satisfactory Stent Placement and Cannula Out
Time Frame: up to 1 hour
Population: Participants/eyes evaluable for primary and secondary outcome measure analysis
Measure: Mean (Standard Deviation); unit: minutes
Units Other Than Participants: Eyes
Groups:
- Conventional Microscope: Conventional microscope used during micro-stent placement.
- NGENUITY: NGENUITY microscope used during micro-stent placement.
Arm/Group | Conventional Microscope | NGENUITY
Number analyzed (Participants) | 13 | 15
Number analyzed (Eyes) | 13 | 16
minutes | 2.55 (1.36) | 3.06 (2.17)
Statistical Analysis 1: Comparison: Conventional Microscope vs NGENUITY; Test type: Other; p = 0.45490734, t-test, 2 sided — The a priori threshold for statistical significance after Bonferroni correction is < 0.002083333

2. Secondary Outcome: Number of Trabecular Meshwork Piercing Attempts Needed to Place Stent
Time Frame: up to 1 hour
Population: Participants/eyes evaluable for primary and secondary outcome measure analysis
Measure: Mean (Standard Deviation); unit: piercing
Units Other Than Participants: Eyes
Arm/Group | Conventional Microscope | NGENUITY
Number analyzed (Participants) | 13 | 15
Number analyzed (Eyes) | 13 | 16
piercing | 1.50 (0.94) | 1.53 (0.92)
Statistical Analysis 1: Comparison: Conventional Microscope vs NGENUITY; Test type: Other; p = 0.92376110, t-test, 2 sided — The a priori threshold for statistical significance after Bonferroni correction is < 0.002083333

3. Secondary Outcome: Number of Anterior Chamber Entry and Reentry Attempts During Stent Placement
Time Frame: up to 1 hour
Population: Participants/eyes evaluable for primary and secondary outcome measure analysis
Measure: Mean (Standard Deviation); unit: Number of Anterior Chamber Entries
Units Other Than Participants: Eyes
Arm/Group | Conventional Microscope | NGENUITY
Number analyzed (Participants) | 13 | 15
Number analyzed (Eyes) | 13 | 16
Number of Anterior Chamber Entries | 1.14 (0.36) | 1.13 (0.35)
Statistical Analysis 1: Comparison: Conventional Microscope vs NGENUITY; Test type: Other; p = 0.94342221, t-test, 2 sided — The a priori threshold for statistical significance after Bonferroni correction is < 0.002083333

4. Secondary Outcome: Number of Microscope Focus or Position Readjustments Needed During Stent Placement
Time Frame: up to 1 hour
Population: Participants/eyes evaluable for primary and secondary outcome measure analysis
Measure: Mean (Standard Deviation); unit: Number of Focus/Microscope adjustments
Units Other Than Participants: Eyes
Arm/Group | Conventional Microscope | NGENUITY
Number analyzed (Participants) | 13 | 15
Number analyzed (Eyes) | 15 | 16
Number of Focus/Microscope adjustments | 1.43 (1.28) | 1.93 (1.79)
Statistical Analysis 1: Comparison: Conventional Microscope vs NGENUITY; Test type: Other; p = 0.38902793, t-test, 2 sided — The a priori threshold for statistical significance after Bonferroni correction is < 0.002083333

5. Secondary Outcome: Change in Attending Questionnaire Score
Description: Providers rate their comfort, visibility, image quality, focus, depth perception, staff engagement, teaching and level of confidence in using the system and system performance. Ratings are on a Likert scale of 1 to 5. Higher scores correspond to excellent ratings, higher confidence in using the system, and better system performance; for Scope Preference only, lower numbers (either group) correspond to a preference for NGenuity visualization.
Time Frame: Up to 5 minutes
Population: Participants/eyes evaluable for primary and secondary outcome measure analysis
Measure: Mean (Standard Deviation); unit: score on a scale
Units Other Than Participants: Eyes
Arm/Group | Conventional Microscope | NGENUITY
Number analyzed (Participants) | 13 | 15
Number analyzed (Eyes) | 13 | 16
score on a scale
  Comfort | 3.14 (0.53) | 3.93 (0.80)
  Visibility | 3.57 (0.85) | 4.53 (0.64)
  Image Quality | 3.14 (0.77) | 4.6 (0.74)
  Focus | 3.14 (0.66) | 4.0 (1.25)
  Depth Perception | 2.93 (0.73) | 4.67 (0.62)
  Staff Engagement | 3.36 (0.50) | 4.27 (0.80)
  Teaching | 3.29 (0.73) | 4.67 (0.62)
  En Face Confidence | 3.43 (0.51) | 4.07 (0.96)
  Hydrus Placement Confidence | 3.71 (0.47) | 4.20 (1.08)
  Scope Preference (1 = 3D.) | 2.71 (0.61) | 1.80 (0.86)
Statistical Analysis 1: Comparison: Conventional Microscope vs NGENUITY; Analysis of comfort score; Test type: Other; p = 0.00424940, t-test, 2 sided — The a priori threshold for statistical significance after Bonferroni correction is < 0.002083333
Statistical Analysis 2: Comparison: Conventional Microscope vs NGENUITY; Analysis of Visibility score; Test type: Other; p = .00223547, t-test, 2 sided — The a priori threshold for statistical significance after Bonferroni correction is < 0.002083333
Statistical Analysis 3: Comparison: Conventional Microscope vs NGENUITY; Analysis of Image Quality score; Test type: Other; p = .00001858, t-test, 2 sided — The a priori threshold for statistical significance after Bonferroni correction is < 0.002083333
Statistical Analysis 4: Comparison: Conventional Microscope vs NGENUITY; Analysis of Focus score; Test type: Other; p = .03003194, t-test, 2 sided — The a priori threshold for statistical significance after Bonferroni correction is < 0.002083333
Statistical Analysis 5: Comparison: Conventional Microscope vs NGENUITY; Analysis of Depth Perception score; Test type: Other; p = .00000028, t-test, 2 sided — The a priori threshold for statistical significance after Bonferroni correction is < 0.002083333
Statistical Analysis 6: Comparison: Conventional Microscope vs NGENUITY; Analysis of Staff Engagement score; Test type: Other; p = .00112148, t-test, 2 sided — The a priori threshold for statistical significance after Bonferroni correction is < 0.002083333
Statistical Analysis 7: Comparison: Conventional Microscope vs NGENUITY; Analysis of Teaching score; Test type: Other; p = 00000951, t-test, 2 sided — The a priori threshold for statistical significance after Bonferroni correction is < 0.002083333
Statistical Analysis 8: Comparison: Conventional Microscope vs NGENUITY; Analysis of En Face Confidence score; Test type: Other; p = .03493564, t-test, 2 sided — The a priori threshold for statistical significance after Bonferroni correction is < 0.002083333
Statistical Analysis 9: Comparison: Conventional Microscope vs NGENUITY; Analysis of Hydrus Placement Confidence score; Test type: Other; p = .12895248, t-test, 2 sided — The a priori threshold for statistical significance after Bonferroni correction is < 0.002083333
Statistical Analysis 10: Comparison: Conventional Microscope vs NGENUITY; Analysis of Scope Preference score; Test type: Other; p = .00279611, t-test, 2 sided — The a priori threshold for statistical significance after Bonferroni correction is < 0.002083333

6. Secondary Outcome: Change in Fellow Questionnaire Score
Description: as for outcome 5
Time Frame: Up to 5 minutes
Population: Participants/eyes evaluable for primary and secondary outcome measure analysis
Measure: Mean (Standard Deviation); unit: score on a scale
Units Other Than Participants: Eyes
Arm/Group | Conventional Microscope | NGENUITY
Number analyzed (Participants) | 13 | 15
Number analyzed (Eyes) | 13 | 16
score on a scale
  Comfort | 4.21 (0.89) | 4.20 (0.56)
  Visibility | 4.21 (0.80) | 4.60 (0.83)
  Image Quality | 4.21 (0.80) | 4.60 (0.83)
  Focus | 3.93 (0.83) | 4.40 (0.91)
  Depth Perception | 4.29 (0.61) | 4.73 (0.59)
  Staff Engagement | 3.57 (0.94) | 4.73 (0.59)
  Teaching | 4.00 (0.78) | 4.80 (0.56)
  En Face Confidence | 4.00 (0.88) | 4.33 (0.82)
  Hydrus Placement Confidence | 4.29 (0.61) | 4.53 (0.83)
  Scope Preference (1 = 3D..) | 3.00 (1.11) | 1.93 (1.10)
Statistical Analysis 1: Comparison: Conventional Microscope vs NGENUITY; Analysis of Comfort score; Test type: Other; p = .959638658, t-test, 2 sided — The a priori threshold for statistical significance after Bonferroni correction is < 0.002083333
Statistical Analysis 2: Comparison: Conventional Microscope vs NGENUITY; Analysis of Visibility score; Test type: Other; p = .213464715, t-test, 2 sided — The a priori threshold for statistical significance after Bonferroni correction is < 0.002083333
Statistical Analysis 3: Comparison: Conventional Microscope vs NGENUITY; Analysis of Image Quality score; Test type: Other; p = .213464715, t-test, 2 sided — The a priori threshold for statistical significance after Bonferroni correction is < 0.002083333
Statistical Analysis 4: Comparison: Conventional Microscope vs NGENUITY; Analysis of Focus score; Test type: Other; p = .155899777, t-test, 2 sided — The a priori threshold for statistical significance after Bonferroni correction is < 0.002083333
Statistical Analysis 5: Comparison: Conventional Microscope vs NGENUITY; Analysis of Depth Perception score; Test type: Other; p = .055960023, t-test, 2 sided — The a priori threshold for statistical significance after Bonferroni correction is < 0.002083333
Statistical Analysis 6: Comparison: Conventional Microscope vs NGENUITY; Analysis of Staff Engagement score; Test type: Other; p = .000685499, t-test, 2 sided — The a priori threshold for statistical significance after Bonferroni correction is < 0.002083333
Statistical Analysis 7: Comparison: Conventional Microscope vs NGENUITY; Analysis of Teaching score; Test type: Other; p = .004526118, t-test, 2 sided — The a priori threshold for statistical significance after Bonferroni correction is < 0.002083333
Statistical Analysis 8: Comparison: Conventional Microscope vs NGENUITY; Analysis of En Face Confidence score; Test type: Other; p = .299921137, t-test, 2 sided — The a priori threshold for statistical significance after Bonferroni correction is < 0.002083333
Statistical Analysis 9: Comparison: Conventional Microscope vs NGENUITY; Analysis of Hydrus Placement Confidence score; Test type: Other; p = .368082084, t-test, 2 sided — The a priori threshold for statistical significance after Bonferroni correction is < 0.002083333
Statistical Analysis 10: Comparison: Conventional Microscope vs NGENUITY; Analysis of Scope Preference score; Test type: Other; p = .015036417, t-test, 2 sided — The a priori threshold for statistical significance after Bonferroni correction is < 0.002083333

ADVERSE EVENTS:
Time Frame: 1 month
Arm/Group | Conventional Microscope | NGENUITY | Conventional Microscope (Re-randomized) | NGENUITY (Re-randomized)
All-Cause Mortality (participants affected / at risk) | 0/14 | 0/14 | 0/1 | 0/3
Serious Adverse Events (participants affected / at risk) | 0/14 | 0/14 | 0/1 | 0/3
Other Adverse Events (participants affected / at risk) | 0/14 | 0/14 | 0/1 | 0/3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2022-10-04): https://cdn.clinicaltrials.gov/large-docs/66/NCT05529966/Prot_000.pdf
  • Statistical Analysis Plan (2025-03-14): https://cdn.clinicaltrials.gov/large-docs/66/NCT05529966/SAP_001.pdf